CLINICAL TRIAL: NCT00751465
Title: Clinical Specificity of Dysfunctional Habitual Attention Processes in Fear of Blushing and Their Changeability
Brief Title: Dysfunctional Attention Processes in Fear of Blushing: Specificity and Changeability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Samia Chaker, Dipl.-Psych., Technische Universität Dresden
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: EK198082007; DFG HO1900/5-1 (Other Grant/Funding Number: Deutsche Forschungsgemeinschaft DFG HO1900/5-1)
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Phobia, Social
Keywords: Social Anxiety Disorder; Social Phobia; Fear of blushing; attention; attention training; cognitive behavior therapy
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Task Concentration Training (Active Comparator): Task Concentration Training TCT following Bögels et al. (1997)
  Interventions: Behavioral: Task Concentration Training
- Standard CBT (Active Comparator): standard Cognitive Behavior Therapy, standard CBT following the model of Clark and Wells (1995).
  Interventions: Behavioral: Standard CBT
- Wait list control (No Intervention): Wait list control group

INTERVENTIONS:
Behavioral: Task Concentration Training — Task Concentration Training TCT following Bögels et al. (1997).
  Arms: Task Concentration Training
Behavioral: Standard CBT — Standard CBT following the Clark-and-Wells (1995) model of social anxiety disorder, relying on the German manual for SAD (stangier et al., 2006). Includes the model, role-plays with and without safetey behavior, video-feedback.
  Arms: Standard CBT

SUMMARY:
Blushing is associated with a heightened self-focused attention. In our study we are interested if this self-focused attention can be shown experimentally and if it can be changed by therapy and training. For the experimental part of the study, we want to compare blushing fearful individuals to social anxious participants who are not fearful of blushing and to healthy controls who report to blush either seldom or quite often. In the therapeutical part of our study, we compare an attention training to the standard cognitive behavioral therapy for social anxiety disorder in an intensive group therapy approach.

DETAILED DESCRIPTION:
Fear of blushing is a specific syndrome in social anxiety disorder. Although attentional biases for social anxiety disorders have often been reported, specific data for fear of blushing are still missing. In this study, dysfunctional attention processes are examined by the use of various questionnaire measures and attention tests (e.g. Stroop test, task switching paradigm) comparing fear of blushers, other social phobia patients, healthy volunteers who report to blush seldomly respectively often. The second goal of the study is to examine if these attention processes can be changed by training and therapy. Therefore, individuals who fulfill DSM-IV criteria for social anxiety disorder and report fear of blushing as main problem, are treated with attention training and with CBT for social anxiety disorder. Therapy will be held in the form of intensive weekend group therapy. Differences in outcomes for both therapy types and in changeability of attention processes on objective test data are examined. Stability of results are tested up to 6-month and 12-month after post-assessment.

ELIGIBILITY:
Inclusion Criteria:

* Social anxiety disorder (DSM-IV criteria) and fear of blushing as main complaint
* age: 18-70

Exclusion Criteria:

* acute severe depression or bipolar disorder
* any disorder of ICD group F2
* acute and severe substance misuse
* any bodily illness which hinders from study participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2008-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Brief Social Phobia Scale | pre, within, post, 6-months, and 12-months follow-up
  Brief Social Phobia Scale BSPS is an interview assessing fear and avoidance in seven social situations and severity of four bodily symptoms.

SECONDARY OUTCOMES:
Social Phobia Composite | pre, within, post, 6-months, and 12-months follow-up
  The social phobia composite includes several self-report measures like the Liebowitz Social Anxiety Scale, Social Phobia Scale, Social Interaction Anxiety Scale, and Social Phobia Inventory.
Changes in objective attention test data | within, post, 6-months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Hoyer, Prof. Dr., Principal Investigator — University of Technology Dresden
Locations (1):
- TU Dresden, Dresden, Germany

REFERENCES:
- [Background] Chaker S, Hofmann SG, Hoyer J. Can a one-weekend group therapy reduce fear of blushing? Results of an open trial. Anxiety Stress Coping. 2010 May;23(3):303-18. doi: 10.1080/10615800903075132. PMID 19557558